CLINICAL TRIAL: NCT00125177
Title: Office for Research on Women's Health (ORWH): Specialized Centers of Research (SCOR) on Sex and Gender Factors Affecting Women's Health. Project 3: Selection Criteria For Muscle Therapy in SUI
Brief Title: IRIS: Incontinence Research Intervention Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P50HD044406 (NIH); 1P50HD044406 (NIH); IRBMED# 2002-0635 (Other: University of Michigan IRB)
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2005-07

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Stress
Keywords: pelvic muscle therapy; urinary incontinence therapy; stress incontinence intervention; incontinence intervention; Incontinence; SUI; Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

INTERVENTIONS:
Behavioral: Knack therapy

SUMMARY:
The IRIS project stands for Incontinence Research Intervention Study. The purpose of this research project is to develop an effective behavioral therapy for urinary incontinence and specifically to test Knack therapy, a self-help treatment. The Knack therapy involves learning the skill of performing a pelvic muscle contraction simultaneously with an event known to trigger leakage, in order to stop that leakage.

DETAILED DESCRIPTION:
This proposal aims to develop and test, in a general population of women with stress urinary incontinence (SUI), a model for predicting who will succeed in overcoming incontinence long-term (1-year) by simply using Knack therapy (thus avoiding invasive and costly surgery and time consuming Kegel's exercises). Specific Aims are to:

* develop a logistic regression model to predict success with the Knack;
* validate the model by determining the proportion of people who succeed according to who is predicted to succeed; and
* develop long-term effectiveness of the Knack (1-year).

The project will be implemented in three phases: model development (n=160 women), model validation (n~160), and long-term follow-up of women who demonstrate response. This will be evaluated immediately and at 1 month and at 3-months and 1-year.

ELIGIBILITY:
Inclusion Criteria:

* Women who are incontinent
* Women who experience leakage with coughing, sneezing or exercising
* Women who are generally healthy
* Women who are over the age of eighteen
* Women who are not pregnant nor expecting to become pregnant within a year

Exclusion Criteria:

* No urine leakage when coughing, sneezing, or exercising
* Under the age of eighteen
* Pregnant or expecting to become pregnant
* Untreated urinary tract infection
* Pronounced pain or discomfort with pelvic exams
* History of neurologic conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2003-01; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The short-term outcome of "positive response" is defined as able to reduce leakage during coughing to under 2 ml or 50% decrease from baseline (whichever is more stringent). This will be evaluated immediately at 1 month.

SECONDARY OUTCOMES:
Long-term success (3-months and 1-year) is defined both by the paper towel test criteria and by documentation of at least 50% reduction of leakage in diary to reflect success at home.

CONTACTS AND LOCATIONS:
Overall Officials: Janis M Miller, PhD, APRN, Principal Investigator — University of Michigan, School of Nursing, Dept. Obstetrics & Gynecology; John OL DeLancey, MD, Study Director — University of Michigan, Obstetrics & Gynecology
Locations (1):
- University of Michigan, School of Nursing, Ann Arbor, Michigan, United States